CLINICAL TRIAL: NCT03729011
Title: Delirium Reduction by Volatile Anesthesia in Cardiac Surgery: Prospective, Randomized, Single-blinded Study
Brief Title: Delirium Reduction by Volatile Anesthesia in Cardiac Surgery
Acronym: DELICATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18
Record Dates: First submitted 2018-10-03; First posted 2018-11-02 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-01

CONDITIONS: Delirium
Keywords: delirium; Cardiac surgery; Cardiopulmonary bypass; Cognitive dysfunction
MeSH Terms: conditions — Delirium; Cognitive Dysfunction | interventions — Sevoflurane; Desflurane; Isoflurane; Propofol

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated to receive either inhalation anaesthesia or TIVA. Permuted-block randomization will be used to allocate subjects to one of the study groups. Sequentially numbered sealed opaque envelopes will contain the treatment code, to be opened in the morning of surgery. Patients will be unaware of group assignment. All the statistical analyses will be performed by the biostatistician not involved in treatment allocation.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Volatile anesthesia group (Active Comparator)
  Interventions: Drug: Volatile agent
- TIVA group (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Volatile agent — Patients will receive volatile agent to provide general anaesthesia, including CPB period. Volatile agents will be administered from anesthesia induction to the end of surgery. Concentration (MAC) of volatile agent will be selected by anaesthesiologist according to clinical situation and patient features.
  Other Names: Sevoflurane; Desflurane; Isoflurane
  Arms: Volatile anesthesia group
Drug: Propofol — Patients will receive propofol and no volatile agent. Propofol will be used for induction and maintenance of anesthesia.
  Arms: TIVA group

SUMMARY:
Parallel group, prospective, randomized, controlled, single-blinded trial. The aim of our study is to test the hypothesis that volatile anesthesia would reduce the incidence of early postoperative delirium in patients undergoing cardiac surgery with CPB as compared to TIVA.

DETAILED DESCRIPTION:
Delirium is a common neurologic complication after cardiac surgery. Up to 52% of postoperative cardiac surgery patients have delirium. The occurrence of postoperative delirium is associated with worse outcomes, including prolonged length of stay in the ICU and hospital, increased morbidity and mortality, compromised long-term cognitive function and physical ability, and elevated medical care costs. Morbidity of postoperative cognitive dysfunction and delirium mostly common in patients with age more than 60 years.

Several factors including cerebral anoxia, embolism, excessive excitatory neurotransmitter release, systemic inflammatory response, electrolyte and metabolic disorders and hemodynamic changes have been demonstrated to contribute to postoperative neurological dysfunction and delirium.

Previous studies have shown that inhalation anaesthesia and total intravenous anaesthesia (TIVA) may produce different degrees of cerebral protection in these patients. Effects of this two types of anaesthesia in cardiac surgery with CPB remain controversial and much debated.

Inhalation agents depress glucose metabolism, decrease cerebral metabolic rate and oxygen consumption. They also partially uncouple the reactivity of cerebral blood flow to CO2. The changes in cerebral blood flow (CBF) depend on the changes in cerebral metabolism and on direct vasodilatory effects. Cerebral autoregulation is dose-dependently altered. Volatile anaesthetics have been shown to initiate early ischemic preconditioning in neurons, but models of focal brain ischemia suggest it can take 24 h for preconditioning to develop fully.

Propofol is a well-known potentiator of GABAA receptors, it reduces cerebrovascular resistance, CBF and cerebral oxygen delivery during cardiopulmonary bypass. A neuroprotective effect of propofol has been shown to be present in many in vitro and in vivo established experimental models of mild/moderate acute cerebral ischemia.

In recent meta-analysis of 13 randomized controlled studies Chen et al compared the neuroprotective effects of inhalational anesthesia and those of total intravenous anesthesia (TIVA) in cardiac surgery with cardiopulmonary bypass. They have shown that anesthesia with volatile agents appeared to provide better cerebral protection than TIVA. As this meta-analysis had several limitations (small sample size of included studies, high heterogenity, etc.), further studies with larger clinically relevant sample-sizes are needed to demonstrate which anesthetics are more beneficial in terms of brain protection in cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Males and females > 65 years
* Written informed consent
* Cardiac surgery with CPB

Exclusion Criteria:

* Emergency surgery
* Surgery on aorta
* Known allergy to components of anaesthesia
* Pregnancy
* Hemodynamically significant stenosis of carotid arteries
* Parkinson's disease
* Liver cirrhosis (Child B or C)
* Current enrollment into another RCT (in the last 30 days)
* Previous enrollment and randomization into the DELICATE trial
* Poor language comprehension
* Preoperative Medications: Anticholinergics (dimedrol, atropine, dramina), antidepressants, antiepileptics, antiparkinson drugs, chemotherapeutic agents

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 405 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Postoperative delirium | 5 days after surgery
  Postoperative delirium detection will be managed with Confusion Assessment Method for the ICU (CAM-ICU)

SECONDARY OUTCOMES:
Early postoperative cognitive dysfunction | 7 days after surgery
  We will use Montreal Cognitive Assessment (MoCA) to detect cognitive dysfunction
Delirium duration | 10 days after surgery
  number of days
Duration of ICU stay | 30 days
  number of days
Duration of hospital stay | 60 days
  number of days
30-day all-cause mortality | 30 days
  yes/no
One-year all-cause mortality | 1 year
  yes/no
Myocardial infarction (MI) | 30 days
  yes/no
Stroke | 30 days
  Stroke will be diagnosed by neurologist (yes/no)
Seizures | 30 days
  Presence of Seizures (yes/no)
Incidence of acute kidney injury (AKI) | 30 days
  According to KDIGO criteria
Renal replacement therapy | 30 days
  We will collect data about need of renal replacement therapy (yes/no)
Infectious complications | 30 days
  We will collect data about infectious complications: wound infection, mediastinitis, pneumonia, positive blood culture
Pain assessment with Behavioral Pain Scale (BPS) | 5 days after surgery
  The BPS is an observational pain scale. It has been validated for use in deeply sedated, mechanically ventilated patients. The BPS contains 3 subscales: facial expression, upper limb movements, and compliance with mechanical ventilation. Each subscale is scored from 1 (no response) to 4 (full response). Therefore, BPS scores range from 3 (no pain) to 12 (maximal pain). A BPS score of 6 or higher is considered to reflect unacceptable pain.
Pain assessment with Numerical Rating Scale (NRS) | 5 days after surgery
  A NRS involves asking the patient to rate his or her pain from 0 to 10 (11 point scale) or from 0 to 100 (101 point scale) with the understanding that 0 is equal to no pain and 10 or 100 is equal to worst possible pain.

CONTACTS AND LOCATIONS:
Locations (5):
- Russia (5):
  - National Medical Research Center for Surgery named after A.V. Vishnevsky, Ministry of Health of the Russian Federation, Moscow
  - M.F. Vladimirsky Moscow Regional Research and Clinical Institute (MONIKI), Moscow
  - Meshalkin Research Institute of Pathology of Circulation, Novosibirsk
  - Saint Petersburg State University Hospital, Saint Petersburg
  - Tomsk National Research Medical Center of the Russian Academy of Sciences, Tomsk

REFERENCES:
- [Background] Brown CH. Delirium in the cardiac surgical ICU. Curr Opin Anaesthesiol. 2014 Apr;27(2):117-22. doi: 10.1097/ACO.0000000000000061. PMID 24514034
- [Background] Martin BJ, Buth KJ, Arora RC, Baskett RJ. Delirium: a cause for concern beyond the immediate postoperative period. Ann Thorac Surg. 2012 Apr;93(4):1114-20. doi: 10.1016/j.athoracsur.2011.09.011. Epub 2011 Dec 24. PMID 22200370
- [Background] Gottesman RF, Grega MA, Bailey MM, Pham LD, Zeger SL, Baumgartner WA, Selnes OA, McKhann GM. Delirium after coronary artery bypass graft surgery and late mortality. Ann Neurol. 2010 Mar;67(3):338-44. doi: 10.1002/ana.21899. PMID 20373345
- [Background] Rudolph JL, Inouye SK, Jones RN, Yang FM, Fong TG, Levkoff SE, Marcantonio ER. Delirium: an independent predictor of functional decline after cardiac surgery. J Am Geriatr Soc. 2010 Apr;58(4):643-9. doi: 10.1111/j.1532-5415.2010.02762.x. Epub 2010 Mar 22. PMID 20345866
- [Background] Franco K, Litaker D, Locala J, Bronson D. The cost of delirium in the surgical patient. Psychosomatics. 2001 Jan-Feb;42(1):68-73. doi: 10.1176/appi.psy.42.1.68. PMID 11161124
- [Background] Pisani MA, Kong SY, Kasl SV, Murphy TE, Araujo KL, Van Ness PH. Days of delirium are associated with 1-year mortality in an older intensive care unit population. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1092-7. doi: 10.1164/rccm.200904-0537OC. Epub 2009 Sep 10. PMID 19745202
- [Background] Bickel H, Gradinger R, Kochs E, Forstl H. High risk of cognitive and functional decline after postoperative delirium. A three-year prospective study. Dement Geriatr Cogn Disord. 2008;26(1):26-31. doi: 10.1159/000140804. Epub 2008 Jun 24. PMID 18577850
- [Background] Li YW, Li HJ, Li HJ, Feng Y, Yu Y, Guo XY, Li Y, Zhao BJ, Hu XY, Zuo MZ, Zhang HY, Wang MR, Ji P, Yan XY, Wu YF, Wang DX. Effects of two different anesthesia-analgesia methods on incidence of postoperative delirium in elderly patients undergoing major thoracic and abdominal surgery: study rationale and protocol for a multicenter randomized controlled trial. BMC Anesthesiol. 2015 Oct 13;15:144. doi: 10.1186/s12871-015-0118-5. PMID 26459347
- [Background] Nguyen Q, Uminski K, Hiebert BM, Tangri N, Arora RC. Midterm outcomes after postoperative delirium on cognition and mood in patients after cardiac surgery. J Thorac Cardiovasc Surg. 2018 Feb;155(2):660-667.e2. doi: 10.1016/j.jtcvs.2017.09.131. Epub 2017 Oct 20. PMID 29132782
- [Background] Cerejeira J, Firmino H, Vaz-Serra A, Mukaetova-Ladinska EB. The neuroinflammatory hypothesis of delirium. Acta Neuropathol. 2010 Jun;119(6):737-54. doi: 10.1007/s00401-010-0674-1. Epub 2010 Mar 24. PMID 20309566
- [Background] Caplan JP, Chang G. Refeeding syndrome as an iatrogenic cause of delirium: a retrospective pilot study. Psychosomatics. 2010 Sep-Oct;51(5):419-24. doi: 10.1176/appi.psy.51.5.419. PMID 20833941
- [Background] Siepe M, Pfeiffer T, Gieringer A, Zemann S, Benk C, Schlensak C, Beyersdorf F. Increased systemic perfusion pressure during cardiopulmonary bypass is associated with less early postoperative cognitive dysfunction and delirium. Eur J Cardiothorac Surg. 2011 Jul;40(1):200-7. doi: 10.1016/j.ejcts.2010.11.024. Epub 2010 Dec 18. PMID 21168339
- [Background] Hshieh TT, Fong TG, Marcantonio ER, Inouye SK. Cholinergic deficiency hypothesis in delirium: a synthesis of current evidence. J Gerontol A Biol Sci Med Sci. 2008 Jul;63(7):764-72. doi: 10.1093/gerona/63.7.764. PMID 18693233
- [Background] Wimmer-Greinecker G, Matheis G, Brieden M, Dietrich M, Oremek G, Westphal K, Winkelmann BR, Moritz A. Neuropsychological changes after cardiopulmonary bypass for coronary artery bypass grafting. Thorac Cardiovasc Surg. 1998 Aug;46(4):207-12. doi: 10.1055/s-2007-1010226. PMID 9776494
- [Background] Chen F, Duan G, Wu Z, Zuo Z, Li H. Comparison of the cerebroprotective effect of inhalation anaesthesia and total intravenous anaesthesia in patients undergoing cardiac surgery with cardiopulmonary bypass: a systematic review and meta-analysis. BMJ Open. 2017 Oct 11;7(10):e014629. doi: 10.1136/bmjopen-2016-014629. PMID 29025825
- [Background] Morimoto Y, Yoshimura M, Utada K, Setoyama K, Matsumoto M, Sakabe T. Prediction of postoperative delirium after abdominal surgery in the elderly. J Anesth. 2009;23(1):51-6. doi: 10.1007/s00540-008-0688-1. Epub 2009 Feb 22. PMID 19234823
- [Background] Sagara Y, Hendler S, Khoh-Reiter S, Gillenwater G, Carlo D, Schubert D, Chang J. Propofol hemisuccinate protects neuronal cells from oxidative injury. J Neurochem. 1999 Dec;73(6):2524-30. doi: 10.1046/j.1471-4159.1999.0732524.x. PMID 10582614
- [Background] Wang H, Lu S, Yu Q, Liang W, Gao H, Li P, Gan Y, Chen J, Gao Y. Sevoflurane preconditioning confers neuroprotection via anti-inflammatory effects. Front Biosci (Elite Ed). 2011 Jan 1;3(2):604-15. doi: 10.2741/e273. PMID 21196338
- [Background] McAuliffe JJ, Loepke AW, Miles L, Joseph B, Hughes E, Vorhees CV. Desflurane, isoflurane, and sevoflurane provide limited neuroprotection against neonatal hypoxia-ischemia in a delayed preconditioning paradigm. Anesthesiology. 2009 Sep;111(3):533-46. doi: 10.1097/ALN.0b013e3181b060d3. PMID 19672176
- [Background] Bilotta F, Stazi E, Zlotnik A, Gruenbaum SE, Rosa G. Neuroprotective effects of intravenous anesthetics: a new critical perspective. Curr Pharm Des. 2014;20(34):5469-75. doi: 10.2174/1381612820666140325110113. PMID 24669972
- [Background] Young Y, Menon DK, Tisavipat N, Matta BF, Jones JG. Propofol neuroprotection in a rat model of ischaemia reperfusion injury. Eur J Anaesthesiol. 1997 May;14(3):320-6. doi: 10.1046/j.1365-2346.1997.00130.x. PMID 9202922
- [Background] Ergun R, Akdemir G, Sen S, Tasci A, Ergungor F. Neuroprotective effects of propofol following global cerebral ischemia in rats. Neurosurg Rev. 2002 Mar;25(1-2):95-8. doi: 10.1007/s101430100171. PMID 11954772
- [Background] Van Aken H, Van Hemelrijck J. Influence of anesthesia on cerebral blood flow and cerebral metabolism: an overview. Agressologie. 1991;32(6-7):303-6. PMID 1843831
- [Background] Lingehall HC, Smulter NS, Lindahl E, Lindkvist M, Engstrom KG, Gustafson YG, Olofsson B. Preoperative Cognitive Performance and Postoperative Delirium Are Independently Associated With Future Dementia in Older People Who Have Undergone Cardiac Surgery: A Longitudinal Cohort Study. Crit Care Med. 2017 Aug;45(8):1295-1303. doi: 10.1097/CCM.0000000000002483. PMID 28481752